CLINICAL TRIAL: NCT01013714
Title: Prophylactic Cardiac Sympathetic Denervation for Prevention of Ventricular Tachyarrhythmias (PREVENT VT)
Brief Title: Cardiac Sympathetic Denervation for Prevention of Ventricular Tachyarrhythmias
Acronym: PREVENT VT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Marmar Vaseghi, Associate Professor of Medicine/Cardiology, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCLA09-07-100-01
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Sudden Cardiac Death; Ventricular Tachycardia; Ventricular Fibrillation; Cardiomyopathy
Keywords: Sudden cardiac death; Ventricular tachycardia; Ventricular fibrillation; Cardiomyopathy; Internal cardiac defibrillator shocks; Internal cardiac defibrillator therapies
MeSH Terms: conditions — Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation; Cardiomyopathies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care + Cardiac Sympathetic Denervation (CSD) (Active Comparator): Patients in this arm receive routine care and undergo cardiac sympathetic denervation. The procedure must be scheduled to occur within one month of randomization.
  Follow-up Visits
  * Follow up at 4 weeks after optimization of medical therapy and surgery
  * All patients are followed at the ICD clinic at 7 months or as needed.
  * Information regarding ICD therapy and arrhythmias will be obtained from ICD interrogations at the follow up visits.
  * Monthly phone calls will be used to determine for interval events, including presence of side-effects.
  VT Ablation is permitted in both arms for ICD shock after optimization.
  Interventions: Procedure: Cardiac Sympathetic Denervation (CSD); Drug: Routine Care
- Routine Care (Placebo Comparator): Patients in this arm remain on prescribed drug regimen and will not undergo CSD.
  Follow-up Visits
  * Medical follow up at 4 weeks after optimization of medical therapy.
  * All patients are followed at the ICD clinic at 7 months or as needed.
  * Information regarding ICD therapy and arrhythmias will be obtained from ICD interrogations at the follow up visits.
  * Monthly phone calls will be used to determine for interval events, including presence of side-effects.
  VT Ablation is permitted in both arms for ICD shock after optimization.
  Interventions: Drug: Routine Care

INTERVENTIONS:
Procedure: Cardiac Sympathetic Denervation (CSD) — Cardiac sympathetic denervation is performed using an endoscopic procedure called VATS (video-assisted thoracoscopic sympathectomy). The surgeon removes the lower half of the stellate ganglia in addition to the thoracic ganglia of T2 - T4 on both the right and left side. The VATS procedure provides a minimally invasive endoscopic approach that is safe and effective. The procedure can be completed in less than 45 minutes on each side.
  Arms: Routine Care + Cardiac Sympathetic Denervation (CSD)
Drug: Routine Care — Anti-arrhythmic medications are continued for the duration of the study unless discontinued or adjusted to due to drug toxicity, intolerance, or ICD shock. All anti-arrhythmic medications (whether in the routine care or surgical arm) can be adjusted at the discretion of the treating physician.

SUMMARY:
The purpose of this research study is to examine the effect of cardiac sympathetic denervation (CSD) surgery on life threatening abnormal heart rhythms called ventricular tachycardia or ventricular fibrillation that can lead to sudden cardiac death. Subjects will be asked to participate in this research study if they have recurrent ventricular tachycardia (at least one ICD shock for ventricular tachycardia) and have undergone at least one catheter ablation procedure or have ventricular tachycardia or fibrillation that is not ablatable. The goal of this study is to determine whether cardiac sympathetic denervation can prevent these abnormal heart rhythms from occurring and therefore, prevent, ICD shocks which are not only painful, but have been shown to reduce quality of life and/or lead to depression, particularly in the period immediately after the shock.

DETAILED DESCRIPTION:
The purpose of this study is to determine if bilateral cardiac sympathetic denervation (CSD) in addition to routine care is more effective than routine care for the treatment of ventricular tachycardia or fibrillation in patients with implantable cardioverter defibrillators (ICDs) who continue to have episodes of VT despite drug therapy and when appropriate, at least one catheter ablation procedure.

The CSD procedure involves removal of part of the cervical stellate ganglia and thoracic ganglia of level 2 to 4. These ganglia house the left and right sided nerves that feed the heart and have been implicated in the occurrence of fast abnormal rhythms that cause defibrillator shocks and sudden death. Stimulation of these nerves has been shown to increase the incidence of sudden death and fast abnormal heart rhythms that lead to internal defibrillator shocks called ventricular tachycardia/ventricular fibrillation. Removal of the ganglia of these nerves in animal and human studies has been shown to decrease the incidence of life threatening abnormal rhythms and sudden death.The procedure takes less than 45 minutes on each side and can be performed endoscopically.

We are inviting patients to participate in this clinical trial who have undergone at least one catheter ablation procedure for ventricular tachycardia but have continued to experience recurrent arrhythmias (ICD shocks) or who have a type of ventricular tachycardia or fibrillation that can not be treated with catheter ablation procedures. Patients will be randomized in a 1:1 fashion to either routine care + cardiac sympathetic denervation (CSD) or routine care without cardiac sympathetic denervation. We are asking 40 individuals (approximate age range 18-80 years) who continue to experience ICD shocks to participate in this research study but only half these individual will be randomized to cardiac sympathetic denervation (CSD) surgery.

ELIGIBILITY:
INCLUSION CRITERIA

1. Appropriate ICD shock for VT after at least one catheter ablation of VT procedure, OR appropriate ICD shock for VT and underwent electrophysiology study/ablation procedure where the procedure was not successful (i.e. determined that VT comes from an inaccessible location or VT was not inducible and could not be targeted or continued to have inducible VT at the end of the procedure) OR appropriate ICD shock for VT and not a candidate for VT ablation (i.e. patients with presence polymorphic VT or ventricular fibrillation, LV thrombus)).
2. Presence of structural heart disease as defined as EF ≤ 50% or presence of ventricular scar as detected by imaging modalities or electroanatomic mapping, hypertrophic cardiomyopathy, cardiac sarcoidosis, or arrhythmogenic right ventricular cardiomyopathy.
3. Patient is taking at least one anti-arrhythmic drug or has documented intolerance or toxicity to at least one anti-arrhythmic drug.
4. 18 years of age or older at time of enrollment
5. Able and willing to comply with all pre- and follow-up testing and requirements.
6. Provision of signed informed consent and stated willingness to comply with all study procedures for duration of the study.

EXCLUSION CRITERIA

1. Active ongoing cardiac ischemia as assessed by: ECG, cardiac enzymes, symptoms, coronary angiography with evidence of significant epicardial coronary stenosis (>70%), or stress testing. (Note: positive troponin assay due to ICD shocks is not an exclusion criterion).
2. Any medical or non-medical condition likely to prevent completion of trial.
3. Contraindication to cardiac sympathetic denervation (i.e. unlikely to tolerate general anesthesia, single-lung ventilation, severe pulmonary disease, or severe pulmonary hypertension) or previous cardiac sympathetic denervation procedure.
4. Left ventricular assist device or status post orthotopic heart transplantation
5. Severe thrombocytopenia (platelets < 50,000) or Coagulopathy (INR > 2.0) that is not due to medications or a reversible cause.
6. Women who are pregnant (as evidenced by pregnancy test if pre-menopausal).
7. Unable or unwilling to comply with protocol requirements.
8. NYHA class IV heart failure symptoms.
9. Known channelopathy such as long QT syndrome and catecholaminergic polymorphic VT.
10. Clinical VT rate < 150 bpm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to ICD shock, death, or cardiac transplantation | 7 months
  To compare the time to first occurrence of appropriate ICD shock, death or cardiac transplantation in CSD+routine care vs. routine care groups.

SECONDARY OUTCOMES:
Number of ICD shocks | 7 months
  To compare the number of ICD shocks in patients with Routine Care + CSD to Routine Care.
Number of appropriate ICD therapies (including ATPs ) and sustained VT below ICD detection | 7 months
  To compare the number of appropriate ICD therapies and VT episodes below ICD detection in patients with Routine Care + CSD to Routine Care.
Serious adverse events | 7 months
  To assess the occurrence of serious adverse events in patients treated with Routine Care + CSD and Routine Care.
Number and etiology of hospitalizations | 7 months
  Number and etiology of hospitalization will be compared in the control vs. intervention group.
Number of deaths or cardiac transplantations | 7 months
  Number of deaths or cardiac transplantation in both arms of the study will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Marmar Vaseghi, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - UCLA Health, Los Angeles, California
  - OHSU, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with other investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years

REFERENCES:
- [Background] Mahajan A, Moore J, Cesario DA, Shivkumar K. Use of thoracic epidural anesthesia for management of electrical storm: a case report. Heart Rhythm. 2005 Dec;2(12):1359-62. doi: 10.1016/j.hrthm.2005.09.004. No abstract available. PMID 16360091
- [Background] Stephenson EA, Berul CI. Electrophysiological interventions for inherited arrhythmia syndromes. Circulation. 2007 Aug 28;116(9):1062-80. doi: 10.1161/CIRCULATIONAHA.106.655779. No abstract available. PMID 17724272
- [Background] Nademanee K, Taylor R, Bailey WE, Rieders DE, Kosar EM. Treating electrical storm : sympathetic blockade versus advanced cardiac life support-guided therapy. Circulation. 2000 Aug 15;102(7):742-7. doi: 10.1161/01.cir.102.7.742. PMID 10942741
- [Background] Tygesen H, Wettervik C, Claes G, Drott C, Emanuelsson H, Solem J, Lomsky M, Radberg G, Wennerblom B. Long-term effect of endoscopic transthoracic sympathicotomy on heart rate variability and QT dispersion in severe angina pectoris. Int J Cardiol. 1999 Aug 31;70(3):283-92. doi: 10.1016/s0167-5273(99)00101-1. PMID 10501343
- [Background] Schwartz PJ, Priori SG, Cerrone M, Spazzolini C, Odero A, Napolitano C, Bloise R, De Ferrari GM, Klersy C, Moss AJ, Zareba W, Robinson JL, Hall WJ, Brink PA, Toivonen L, Epstein AE, Li C, Hu D. Left cardiac sympathetic denervation in the management of high-risk patients affected by the long-QT syndrome. Circulation. 2004 Apr 20;109(15):1826-33. doi: 10.1161/01.CIR.0000125523.14403.1E. Epub 2004 Mar 29. PMID 15051644
- [Background] Li J, Wang L, Wang J. Video-assisted thoracoscopic sympathectomy for congenital long QT syndromes. Pacing Clin Electrophysiol. 2003 Apr;26(4 Pt 1):870-3. doi: 10.1046/j.1460-9592.2003.t01-1-00152.x. PMID 12715848
- [Background] Ouriel K, Moss AJ. Long QT syndrome: an indication for cervicothoracic sympathectomy. Cardiovasc Surg. 1995 Oct;3(5):475-8. doi: 10.1016/0967-2109(95)94444-2. PMID 8574528
- [Background] Lobato EB, Kern KB, Paige GB, Brown M, Sulek CA. Differential effects of right versus left stellate ganglion block on left ventricular function in humans: an echocardiographic analysis. J Clin Anesth. 2000 Jun;12(4):315-8. doi: 10.1016/s0952-8180(00)00158-6. PMID 10960205
- [Background] Schlack W, Dinter W. Haemodynamic effects of a left stellate ganglion block in ASA I patients. An echocardiographic study. Eur J Anaesthesiol. 2000 Feb;17(2):79-84. doi: 10.1046/j.1365-2346.2000.00606.x. PMID 10758450
- [Background] Bourke T, Vaseghi M, Michowitz Y, Sankhla V, Shah M, Swapna N, Boyle NG, Mahajan A, Narasimhan C, Lokhandwala Y, Shivkumar K. Neuraxial modulation for refractory ventricular arrhythmias: value of thoracic epidural anesthesia and surgical left cardiac sympathetic denervation. Circulation. 2010 Jun 1;121(21):2255-62. doi: 10.1161/CIRCULATIONAHA.109.929703. Epub 2010 May 17. PMID 20479150
- [Background] Ajijola OA, Vaseghi M, Mahajan A, Shivkumar K. Bilateral cardiac sympathetic denervation: why, who and when? Expert Rev Cardiovasc Ther. 2012 Aug;10(8):947-9. doi: 10.1586/erc.12.93. No abstract available. PMID 23030281
- [Background] Johnson JP, Ahn SS, Choi WC, Masciopinto JE, Kim KD, Filler AG, Desalles AA. Thoracoscopic sympathectomy: techniques and outcomes. Neurosurg Focus. 1998 Feb 15;4(2):e4. doi: 10.3171/foc.1998.4.2.7. PMID 17206769
- [Background] Vaseghi M, Gima J, Kanaan C, Ajijola OA, Marmureanu A, Mahajan A, Shivkumar K. Cardiac sympathetic denervation in patients with refractory ventricular arrhythmias or electrical storm: intermediate and long-term follow-up. Heart Rhythm. 2014 Mar;11(3):360-6. doi: 10.1016/j.hrthm.2013.11.028. Epub 2013 Nov 28. PMID 24291775
- [Background] Vaseghi M, Barwad P, Malavassi Corrales FJ, Tandri H, Mathuria N, Shah R, Sorg JM, Gima J, Mandal K, Saenz Morales LC, Lokhandwala Y, Shivkumar K. Cardiac Sympathetic Denervation for Refractory Ventricular Arrhythmias. J Am Coll Cardiol. 2017 Jun 27;69(25):3070-3080. doi: 10.1016/j.jacc.2017.04.035. PMID 28641796